CLINICAL TRIAL: NCT00216359
Title: The Radata-Fuzeon Cohort - An Observational Cohort-Study in HIV-Infected Patients Using Fuzeon (Enfuvirtide) as Part of Their Antiretroviral Combination Therapy
Brief Title: Cohort Study for Patients Using Fuzeon (Enfuvirtide)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institute for Interdisciplinary Infectiology (Other)
Collaborators: Hoffmann-La Roche (Industry)
Other Study IDs: Radata Fuzeon Cohort
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; Antiretroviral Treatment
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

INTERVENTIONS:
Drug: Fuzeon (Enfuvirtide)
Procedure: Laboratory diagnostic (CD4-cells)
Procedure: Laboratory diagnostics (HIV-1 viral load)
Drug: antiretroviral co-medication beside Fuzeon

SUMMARY:
The Radata-Fuzeon cohort is an observational cohort study to gain a better understanding of Fuzeon (Enfuvirtide) in daily clinical practice. Patients planned to take this drug in a new antiretroviral combination therapy (ART) are eligible to participate in this observation.

Physicians may register patients online via the internet. They are offered to get an expert advice suggesting therapeutics for a new ART.

Observation interval is every three month. However physicians are allowed to initiate new diagnostics, expert advice and therapeutic changes independently from these intervals if necessary.

Total observation time for each patients is planned for two years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV-Infection
* Planned to switch to a Fuzeon-containing antiretroviral therapy

Exclusion Criteria:

* Inability to understand or sign inform consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2003-05; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Plettenberg, MD, Study Chair — ifi-Institute for Interdisciplinary Infectiology
Locations (1):
- Ifi-Institute for Interdisciplinary Infectiology, Hamburg, Germany

REFERENCES:
- See also: Radata-Homepage (German language) — http://www.radata.de